CLINICAL TRIAL: NCT04231097
Title: Mindfulness-Based Cognitive Therapy Delivered Via Group Videoconferencing for Acute Coronary Syndrome Patients With Depressive Symptoms
Brief Title: MBCT Delivered Via Group Videoconferencing for ACS Syndrome Patients With Depressive Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Christina Luberto, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020P000045
Record Dates: First submitted 2020-01-10; First posted 2020-01-18 (Actual); Results first posted 2023-04-24 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2023-04

CONDITIONS: Acute Coronary Syndrome; Depression; Myocardial Infarction; Unstable Angina; STEMI; NSTEMI - Non-ST Segment Elevation MI
Keywords: Mindfulness; Acute Coronary Syndrome; Videoconferencing; Depression
MeSH Terms: conditions — Acute Coronary Syndrome; Depression; Myocardial Infarction; Angina, Unstable; ST Elevation Myocardial Infarction; Non-ST Elevated Myocardial Infarction

STUDY DESIGN:
Intervention Model Description: Approximately N=20 patients (2 cohorts of 10 participants/per cohort, accounting for 20% anticipated lost to follow-up). Assignment to each cohort will be based on timing and/or participant scheduling preferences. Intervention cohort groups will be run either concurrently or sequentially, depending on the enrollment frequency of participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Virtual MBCT (Experimental): Two cohorts of MBCT participants with approximately 10 participants per cohort.
  Interventions: Other: MBCT intervention for ACS patients

INTERVENTIONS:
Other: MBCT intervention for ACS patients — The MBCT intervention will involve 8 virtually-delivered MBCT sessions (approximately 1.5 hours each), during which participants will be taught how to use evidence-based mindfulness skills to regulate distress and choose healthy behaviors, as well as learn about cardiac health. Participants involved in the intervention will be asked to complete a brief survey following each session. Within one week before and after the intervention and 3-months post-intervention participants will be asked to complete a series of questionnaires and provide self-collected blood samples. Upon completion of the intervention participants will complete an audio-or video recorded exit interview (approximately 30 minutes).

SUMMARY:
Brief Summary: The aim of this study is to explore the initial feasibility and acceptability of (a) Mindfulness-Based Cognitive Therapy (MBCT) adapted for ACS patients; (b) the group videoconferencing delivery medium; and (c) dried blood spot research procedures, to inform refinements for a subsequent pilot RCT.

DETAILED DESCRIPTION:
The current study will employ an open pilot trial to determine the initial feasibility and acceptability of a targeted, virtual MBCT intervention for ACS patients. The investigators plan to enroll approximately N=20 patients (2 cohorts of 10 participants/per cohort, accounting for 20% anticipated lost to follow-up). The MBCT intervention will involve 8 virtually-delivered MBCT sessions (approximately 1.5 hours each), during which participants will be taught how to use evidence-based mindfulness skills to regulate distress and choose healthy behaviors, as well as learn about cardiac health. Participants will be asked to complete a brief survey following each session. Within one week before and after the intervention and 3-months post-intervention participants will be asked to complete a series of questionnaires and provide self-collected blood samples. Upon completion of the intervention participants will complete an audio-or video recorded exit interview (approximately 30 minutes).

Participants will be recruited through the the hospital's clinical data registry, advertisements (e.g., flyers, brochures) placed throughout the hospital, direct provider referrals, and from inpatient cardiac units. Patients who express interest in the study will be asked complete an eligibility screening. Eligible patients agreeable with study participation will then complete a written consent with study staff prior to enrollment.

Participants will be enrolled in one of two MBCT intervention cohorts and expected to participate in 8-weekly, 1.5-hour virtual sessions, in conjunction with approximately 30 minutes of at-home daily practice. A licensed mental health provider (e.g., LICSW, PhD) trained in the MBCT protocol will deliver the intervention. The MBCT intervention will be delivered Zoom, a secure, HIPPA-compliant video-conferencing software.

Study assessments will include a battery of self-report surveys administered at baseline, post-intervention, and 3-month follow-up; session satisfaction surveys administered after each intervention session; post-intervention individual exit interviews (conducted via telephone or videoconference); blood spot samples self-collected by participants at baseline, post-intervention, and 3-month follow-up (submitted to the research team via paper mail); and home practice logs submitted between each intervention session. Primary outcomes for the intervention are feasibility and acceptability. Data collected from the study will be used to assist in the development of future RCTs.

ELIGIBILITY:
Inclusion Criteria:

1. Lifetime ACS per medical record and/or patient confirmation
2. Current elevated depression symptoms (PHQ-9>5)
3. Age 35-85 years
4. Access to high-speed internet

Exclusion Criteria:

1. Active suicidal ideation or past-year psychiatric hospitalization (per patient report and/or medical record review)
2. Non-English-speaking
3. Cognitive impairments preventing informed consent per medical record review and/or cognitive Screen < 4
4. Patient deemed unable to complete the study protocol or has a condition that would likely interfere with the study

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2020-04-24 (Actual); Primary Completion 2021-02-25 (Actual); Study Completion 2021-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christina Luberto, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Mongan Institute: Health Policy Research Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred from April 2020 - September 2020. Patient were recruited from the study hospital using hospital databases, research invitation letters, provider referrals, and flyers. Patients were also recruited in person while hospitalized.
Pre-assignment Details: There is one intervention arm (MBCT). We enrolled two MBCT cohorts of 2 and 6 people each, totaling 8 people. Data are reported for all enrolled participants.
Groups:
- Virtual MBCT: MBCT intervention for ACS patients: The MBCT intervention will involve 8 virtually-delivered MBCT sessions (approximately 1.5 hours each/week) delivered via group videoconferencing, during which participants will be taught how to use evidence-based mindfulness skills to regulate distress and choose healthy behaviors, as well as learn about cardiac health. Participants involved in the intervention will be asked to complete a brief survey following each session. Within one week before and after the intervention and 3-months post-intervention participants will be asked to complete a series of questionnaires and provide self-collected blood samples. Upon completion of the intervention participants will complete an audio-or video recorded exit interview (approximately 30 minutes).
Period: Overall Study
Arm/Group | Virtual MBCT
Started | 8
Completed | 4
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | Virtual MBCT
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.5 (14.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 1
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Recruitment Feasibility: Percent of Participants Who Consent to Screening
Description: Feasibility outcomes for recruitment will include: >70% of patients reached consent to screening
Time Frame: 6 months
Population: Hospital patients meeting preliminary eligibility criteria for ACS, who were approached and consented for eligibility screening
Measure: Count of Participants; unit: Participants
Arm/Group | Virtual MBCT
Number analyzed (Participants) | 191
Participants | 150

2. Primary Outcome: Recruitment Feasibility: Percent of Participants Meeting Screening Criteria
Description: Feasibility outcomes for recruitment will include: >70% meet screening criteria
Time Frame: 6 months
Population: Percent of hospital patients who met preliminary and eligibility screening criteria for ACS. The number who were reached by phone for eligibility screening is 150, but 96 did not complete the full screening protocol and were removed from subsequent analyses. Thus, there were 54 screening completers. The screening outcome is the number eligible out of the 54 who agreed to be completely screened.
Measure: Count of Participants; unit: Participants
Arm/Group | Virtual MBCT
Number analyzed (Participants) | 54
Participants | 12

3. Primary Outcome: Recruitment Feasibility: Percent of Eligible Patients Who Consent
Description: Feasibility outcomes for recruitment will include: >70% of eligible consent to the study
Time Frame: 6 Months
Population: Percent of hospital patients who met eligibility screening criteria and chose to enroll
Measure: Count of Participants; unit: Participants
Arm/Group | Virtual MBCT
Number analyzed (Participants) | 12
Participants | 8

4. Primary Outcome: MBCT Feasibility: Percent of Participants Adherent to the MBCT Intervention
Description: MBCT feasibility will be measured by: >75% session attendance (i.e., percent who attend at least 6/8 intervention sessions)
Time Frame: 6 Months
Population: percent of ITT participants who attended >6/8 session among those who enrolled
Measure: Count of Participants; unit: Participants
Arm/Group | Virtual MBCT
Number analyzed (Participants) | 8
Participants
  ITT analysis | 4
  Completer analysis: number analyzed (Participants) | 4
  Completer analysis | 4

5. Primary Outcome: MBCT Feasibility: Percent of Participants Retained at Post-Intervention
Description: MBCT feasibility will be measured by: >75% post-intervention assessments completed
Time Frame: 3 Months
Population: >75% post-intervention assessments completed among treatment completers and ITT Sample
Measure: Count of Participants; unit: Participants
Arm/Group | Virtual MBCT
Number analyzed (Participants) | 8
Participants
  ITT analysis | 4
  Completer analysis: number analyzed (Participants) | 4
  Completer analysis | 4

6. Primary Outcome: Videoconferencing Feasibility: Percent of Connections Dropped During Sessions
Description: Videoconferencing feasibility will be assessed by: < 20% of connections dropped during session
Time Frame: 6 Months
Population: percent of connections dropped throughout the 8 sessions for both groups (16 sessions)
Measure: Count of Units; unit: Number of virtual sessions
Units Other Than Participants: Number of virtual sessions
Arm/Group | Virtual MBCT
Number analyzed (Participants) | 8
Number analyzed (Number of virtual sessions) | 16
Number of virtual sessions | 1

7. Primary Outcome: Blood Spot Feasibility: Percent of Participants Submitting Blood Spot Samples at Baseline
Description: Blood spot feasibility will be assessed by: >75% of participants submitting samples at baseline
Time Frame: 6 months
Population: percent of participants who submitted samples at baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Virtual MBCT
Number analyzed (Participants) | 8
Participants
  ITT Sample | 4
  Completers: number analyzed (Participants) | 2
  Completers | 2

8. Primary Outcome: Blood Spot Feasibility: Percent of Participants Submitting Blood Spot Sample at Post-Intervention
Description: Blood spot feasibility will be assessed by: >75% of participants submitting samples at post-intervention
Time Frame: 6 Month
Population: Blood spot feasibility will be assessed by: >75% of participants who submitted samples at post-intervention among Completers and ITT sample
Measure: Count of Participants; unit: Participants
Arm/Group | Virtual MBCT
Number analyzed (Participants) | 8
Participants
  ITT analysis | 4
  Completer analysis: number analyzed (Participants) | 4
  Completer analysis | 4

9. Primary Outcome: Blood Spot Feasibility: Percent of Participants Submitting Blood Spot Samples at Follow-up
Description: Blood spot feasibility will be assessed by: >60% of participants submitting samples at follow-up
Time Frame: 6 Months
Population: Blood spot feasibility will be assessed by: >60% of participants who submitted samples at follow-up among Completers and ITT sample
Measure: Count of Participants; unit: Participants
Arm/Group | Virtual MBCT
Number analyzed (Participants) | 8
Participants
  ITT | 4
  Completers: number analyzed (Participants) | 4
  Completers | 4

10. Primary Outcome: Blood Spot Feasibility: Percent of Adequate Blood Spot Samples Submitted
Description: Blood spot feasibility will be assessed by: 80% of samples of adequate quality for processing.
Time Frame: 6 Months
Population: percent of submitted samples with adequate quality for processing
Measure: Count of Units; unit: Samples submitted for processing
Units Other Than Participants: Samples submitted for processing
Arm/Group | Virtual MBCT
Number analyzed (Participants) | 8
Number analyzed (Samples submitted for processing) | 12
Samples submitted for processing | 9

11. Primary Outcome: MBCT Acceptability: Helpfulness for Mood
Description: Ratings of how helpful the MBCT sessions were for improving mood (1 = not at all helpful to 10 = very helpful), with acceptability defined as Mean >= 7.5
Time Frame: 6 months
Population: Participants who completed at least one intervention session
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Virtual MBCT
Number analyzed (Participants) | 8
units on a scale | 6.98 (1.40)

12. Primary Outcome: MBCT Acceptability: Usefulness of Session Components
Description: The average usefulness ratings for session components on a scale of 1 = not at all useful to 10 = very useful, with mean >= 7.5 being considered acceptable
Time Frame: 6 months
Population: Participants who completed at least one intervention session
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Virtual MBCT
Number analyzed (Participants) | 8
units on a scale | 7.61 (1.55)

13. Primary Outcome: Videoconferencing Acceptability: Ratings of Videoconferencing Ease of Use
Description: Videoconferencing acceptability will be assessed in terms of ease of use (1= very much, 10 = not at all; M >= 7.5)
Time Frame: 6 Months
Population: Average rating for the level of ease of using videoconferencing for intervention sessions throughout the program
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Virtual MBCT
Number analyzed (Participants) | 8
score on a scale | 8.60 (1.60)

14. Primary Outcome: Videoconferencing Acceptability: Ratings of Videoconferencing Quality Surveys)
Description: Videoconferencing acceptability will be assessed in terms of video quality of mindfulness videoconference sessions (1= Very Poor to 10 = Very Good, M>7.5)
Time Frame: 6 Months
Population: Average rating for video quality of mindfulness videoconference sessions through all groups for participants who attended at least one session
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Virtual MBCT
Number analyzed (Participants) | 8
score on a scale | 8.81 (1.42)

15. Primary Outcome: Videoconferencing Acceptability: Ratings of Videoconferencing Satisfaction
Description: Videoconferencing acceptability will be assessed in overall satisfaction of use (1 = not at all satisfied to 10 = very satisfied, M > 7.5)
Time Frame: 6 Months
Population: Average rating for overall satisfaction of videoconferencing for mindfulness sessions across all groups for participants who attended at least one group
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Virtual MBCT
Number analyzed (Participants) | 8
score on a scale | 9.75 (.05)

16. Primary Outcome: Blood Spot Acceptability: Ease of Blood Spot Collection
Description: Blood spot acceptability will be assessed by ratings of ease of blood spot collection (1 = not at all, 10 = very easy; M>7.5)
Time Frame: Average rating for ease of data submission from blood spot collection through out all groups
Population: Blood spot acceptability will be assessed by ratings of ease of blood spot collection
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Virtual MBCT
Number analyzed (Participants) | 8
score on a scale | 7.3 (4.9)

17. Primary Outcome: Blood Spot Acceptability: Discomfort of Blood Spot Collection
Description: Blood spot acceptability will be assessed by ratings of level of pain during blood spot collection, (1=Very much pain, 10=Very little pain; M>=7.5).
Time Frame: 6 Months
Population: Average rating for the level of pain during blood spot collection
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Virtual MBCT
Number analyzed (Participants) | 8
score on a scale | 9.5 (0.58)

18. Secondary Outcome: Patient Health Questionnaire (PHQ-9)
Description: This is a 9-item scale that measures depression. The scoring scale ranges from 0, not at all, to 3, nearly every day. The scoring values range from 0-18, where high values represent higher levels of depression and lower values represent lower levels of depression. Changes of >= 3 points from before to after the intervention represent clinically meaningful change. The outcome is the % of participants who report clinically meaningful change
Time Frame: 6 months
Population: Participants who completed the post-intervention survey with data available for analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Virtual MBCT
Number analyzed (Participants) | 8
Participants | 3

ADVERSE EVENTS:
Time Frame: 6 months from enrollment
Arm/Group | Virtual MBCT
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2020-07-07): https://cdn.clinicaltrials.gov/large-docs/97/NCT04231097/Prot_000.pdf
  • Statistical Analysis Plan (2023-04-04): https://cdn.clinicaltrials.gov/large-docs/97/NCT04231097/SAP_001.pdf
  • Informed Consent Form (2020-12-03): https://cdn.clinicaltrials.gov/large-docs/97/NCT04231097/ICF_002.pdf